CLINICAL TRIAL: NCT00031980
Title: Phase II Study of Cyclosporine in T-Cell Large Granular Lymphocytic Leukemia
Brief Title: Cyclosporine in Treating Patients With Low Blood Counts Caused By Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CALGB-10003; CALGB-10003; CDR0000069246 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Anemia; Leukemia; Neutropenia; Thrombocytopenia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; anemia; neutropenia; thrombocytopenia
MeSH Terms: conditions — Anemia; Leukemia; Neutropenia; Thrombocytopenia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cyclosporine (Experimental): Patients receive oral cyclosporine every 12 hours. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 4 months for 1 year and then every 6 months for 9 years.
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Drug: cyclosporine

SUMMARY:
RATIONALE: Cyclosporine may improve low blood counts caused by hematologic cancer.

PURPOSE: Phase II trial to study the effectiveness of cyclosporine in treating patients who have low blood counts caused by hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of cytopenic response in patients with T-cell large granular lymphocytic leukemia treated with cyclosporine.

OUTLINE: This is a multicenter study.

Patients receive oral cyclosporine every 12 hours. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 4 months for 1 year and then every 6 months for 9 years.

PROJECTED ACCRUAL: A total of 9-30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of T-cell large granular lymphocytic leukemia

  * Increased numbers of large granular lymphocytes in peripheral blood smears
  * CD3+CD8+CD57+ immunophenotype by flow cytometry AND
  * CD3+CD57+ cell count at least 2,000/mm^3 OR
  * CD3+CD57+ cell count at least 500/mm^3 with clonal T-cell receptor beta gene rearrangement
* Patients must have at least 1 of the following:

  * Severe neutropenia (absolute neutrophil count (ANC) less than 500/mm^3)
  * Neutropenia (ANC less than 1,000/mm^3) and recurrent infections
  * Anemia (hemoglobin less than 9 g/dL)
  * Thrombocytopenia (platelet count less than 50,000/mm^3)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* NCI CTC 0-3

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 2 times ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Endocrine therapy:

* No concurrent hormonal therapy except steroids for adrenal failure or hormones for nondisease-related conditions (e.g., insulin for diabetes)
* No concurrent dexamethasone or other steroidal antiemetics

Other:

* No prior cyclosporine therapy for this leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Frequency of cytopemic response | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria R. Baer, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States